CLINICAL TRIAL: NCT05364307
Title: Identification of Mild Cognitive Impairment (MCI) and Early Alzheimer's Disease (AD) Patients With a High Probability of Meeting Eligibility Criteria for a Therapeutic Alzheimer's Disease Clinical Trial (APHELEIA)
Brief Title: Identification of Patients With a High Probability of Meeting Eligibility Criteria for an Alzheimer's Disease Clinical Trial (APHELEIA)
Status: Completed | Type: Observational
Sponsor: Global Alzheimer's Platform Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: Apheleia-001
Record Dates: First submitted 2022-05-04; First posted 2022-05-06 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Memory Loss; Memory Disorders; Memory Impairment
Keywords: Alzheimer's Disease; Memory Loss; Memory Disorder; Mild Cognitive Impairment; Early Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Aβ 42/40, Aβ 42, Aβ40, ApoE4, APS
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prescreener database — Identify and characterize participants with reported memory complaints and/or cognitive impairment to determine the probability of randomization into a therapeutic AD clinical trial.

SUMMARY:
Apheleia-001 is a prescreener that aims to identify and characterize participants with reported cognitive impairment using demographic information, clinical history, brief cognitive assessments, and blood-based biomarkers to distinguish appropriate participants for referral to a therapeutic AD clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants and/or a legally authorized representative (LAR) must provide signed and dated informed consent and authorization to use personal health information in accordance with local and national guidance and regulations;

  2. Male or female 50 to 90 years of age (inclusive) at the time of consent;

  3. Participants must have a Mini-Mental State Exam (MMSE) score of 20 to 28 inclusive;

  4. Progressive cognitive complaints must be reported by participant or caregiver;

  5. Participants must be willing to comply with all procedures as outlined in the informed consent, including blood sampling, genetic testing, and storage of biospecimens for future research;

  6. Fluency in the language of the tests used at the site;

  7. Participants must be interested in participating in clinical research.

Exclusion Criteria:

* 1. Participants who, in the opinion of the Investigator, have serious or unstable medical conditions that would prohibit their completion of all prescreening procedures and data collection;

  2. Participants who are currently enrolled in another clinical study.

  3. Participants who have serious or unstable medical conditions that would likely preclude their participation in an interventional research trial;

  4. Participants who have reported or have a known negative amyloid PET scan in the past 24 months;

  5. Participants with history of stroke within 6 months of prescreening;

  6. Participants with an uncontrolled seizure disorder, unexplained blackouts, OR history of a seizure within 6 months (subjects with a history of pediatric febrile seizure, benign rolandic epilepsy may participate);

  7. Participants with a history or evidence of a malignancy within the 2 years prior to prescreening. Subjects with indolent malignancies (e.g., basal cell carcinoma or squamous cell carcinoma) or malignancies considered to be cured and not actively treated with anti-cancer therapy or radiotherapy are permitted to enroll;

  8. Participants with known or suspected alcohol or drug abuse or dependence within 2 years of prescreening;

  9. Participants with a reported suicidal attempt within 2 years of prescreening), or any unstable psychiatric symptoms (e.g., uncontrolled depression);

  10. Participants who have participated in a clinical trial of any potential disease modifying AD treatment and received active drug within 6 months prior to prescreening;

  11. Participants who have any neurological disorder affecting the central nervous system, other than AD, that may be contributing to cognitive impairment (e.g., Parkinson's disease, other dementias, multiple concussions or seizures) as deemed significant by the Investigator;

  12. Participants with known history of hepatitis C virus, hepatitis B virus, human immunodeficiency virus (HIV) or other immunodeficiencies;

  13. Participants that have previously been consented to this protocol;

  14. Participants with a hypersensitivity to mAb treatments, protein derived from a mAb, or immunoglobulin therapy;

  15. Participants with allergies to diphenhydramine, epinephrine, and methylprednisolone;

  16. Participants who are direct employees or family members of direct employees of the participating investigators' sites;

  17. Participants who are direct employees of the Sponsor;

  18. Participants who, in the opinion of the Investigator, are unable to complete cognitive testing due to inadequate visual or auditory acuity.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 3,000 participants.
Sampling Method: Non-Probability Sample
Enrollment: 1555 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Determine number of patients eligible for therapeutic Alzheimer's Disease clinical trial | Throughout study completion, an average of 45 days
  Participants with reported memory complaints and/or cognitive impairment will provide demographic information, clinical history, complete brief cognitive assessments, and provide blood-based biomarkers

CONTACTS AND LOCATIONS:
Locations (19):
- United States (18):
  - Pacific Research Network, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Visionary Investigator's Network, Aventura, Florida
  - Charter Research, Lady Lake, Florida
  - JEM Research Institute, Lake Worth, Florida
  - ClinCloud, LLC, Maitland, Florida
  - K2 Medical Research, Maitland, Florida
  - Merritt Island Medical Research, Merritt Island, Florida
  - Renstar Medical Research, Ocala, Florida
  - ClinCloud, LLC, Viera, Florida
  - Premiere Research Institute at Palm Beach Neurology, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Charter Research, Winter Park, Florida
  - iResearch, Decatur, Georgia
  - Quest Research Institute, Farmington Hills, Michigan
  - IPS Research, Oklahoma City, Oklahoma
  - Clinical Trials of Texas, San Antonio, Texas
  - Re:Cognition Health, Fairfax, Virginia
- OCT Research, Kelowna, British Colombia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baek MJ, Kim K, Park YH, Kim S. The Validity and Reliability of the Mini-Mental State Examination-2 for Detecting Mild Cognitive Impairment and Alzheimer's Disease in a Korean Population. PLoS One. 2016 Sep 26;11(9):e0163792. doi: 10.1371/journal.pone.0163792. eCollection 2016. PMID 27668883
- [Background] Berry CC. A tutorial on confidence intervals for proportions in diagnostic radiology. AJR Am J Roentgenol. 1990 Mar;154(3):477-80. doi: 10.2214/ajr.154.3.2106207. No abstract available.
- [Background] Jack CR Jr, Bennett DA, Blennow K, Carrillo MC, Dunn B, Haeberlein SB, Holtzman DM, Jagust W, Jessen F, Karlawish J, Liu E, Molinuevo JL, Montine T, Phelps C, Rankin KP, Rowe CC, Scheltens P, Siemers E, Snyder HM, Sperling R; Contributors. NIA-AA Research Framework: Toward a biological definition of Alzheimer's disease. Alzheimers Dement. 2018 Apr;14(4):535-562. doi: 10.1016/j.jalz.2018.02.018. PMID 29653606
- [Background] Kantarci K. Molecular imaging of Alzheimer disease pathology. AJNR Am J Neuroradiol. 2014 Jun;35(6 Suppl):S12-7. doi: 10.3174/ajnr.A3847. Epub 2014 Feb 6. PMID 24503555
- [Background] Niemantsverdriet E, Valckx S, Bjerke M, Engelborghs S. Alzheimer's disease CSF biomarkers: clinical indications and rational use. Acta Neurol Belg. 2017 Sep;117(3):591-602. doi: 10.1007/s13760-017-0816-5. Epub 2017 Jul 27. PMID 28752420
- [Background] O'Bryant SE, Humphreys JD, Smith GE, Ivnik RJ, Graff-Radford NR, Petersen RC, Lucas JA. Detecting dementia with the mini-mental state examination in highly educated individuals. Arch Neurol. 2008 Jul;65(7):963-7. doi: 10.1001/archneur.65.7.963. PMID 18625866